CLINICAL TRIAL: NCT04574674
Title: Effect of a Home-based REsistance Exercise vs a Home-based FLEXbility Exercise Programme on Muscular Endurance and Flexibility in Healthy Adults
Brief Title: Home-based REsistance vs a Home-based FLEXbility Exercise Programmes on Muscular Endurance and Flexibility in Adults
Acronym: REFLEX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Professor Jason Gill, Professor, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200190188
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Exercise
Keywords: muscle endurance; muscle strength; muscular fitness; resistance training; strength training; physical activity; voluntary failure
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial with two groups, flexibility exercise group and resistance exercise group.
Who Masked: Outcomes Assessor
Masking Description: Members of the research team that perform measurements are blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexibility exercise group (Experimental): Participants will be asked to follow a 12-week flexibility exercise training programme. Participants will be asked to perform a minimum amount of flexibility exercise of 1 set/week for each of six exercises and will have the opportunity to increase their volume of exercise to 2 sets or 3 sets/week per exercise if it is their choice.
  Participants will perform 6 flexibility exercises per week (2 different for legs, 1 shoulder and arms, 1 chest, 1 back and 1 core). Passive static stretching exercises will be performed.
  Interventions: Behavioral: Flexibility exercise programme
- Resistance exercise group (Experimental): Participants will be asked to follow a 12-week home-based exercise programme. Participants will be asked to perform a minimum amount of resistance exercise of 1 set/week for each of six exercises and will have the opportunity to increase their volume of exercise to 2 sets or 3 sets/week per exercise if it is their choice.
  Participants in the resistance exercise group will be asked to perform a total of 6 exercises per week (2 different leg exercises, 1 shoulder exercise, 1 chest exercise, 1 back exercise and 1 core exercise). Body weight and resistance bands exercises will be used. Participants will be asked to perform each set to complete as many repetitions as possible until fatigue.
  Interventions: Behavioral: Resistance exercise programme

INTERVENTIONS:
Behavioral: Flexibility exercise programme — Static passive flexibility exercises.
  Arms: Flexibility exercise group
Behavioral: Resistance exercise programme — Body weight and resistance bands exercises.
  Arms: Resistance exercise group

SUMMARY:
This study will evaluate the effects of a home-based resistance exercise programme v/s a home-based flexibility exercise programme on muscular endurance and flexibility on healthy adults. Half of the participants will undergo a 12-weeks home-based resistance exercise programme while the other half will undergo a 12-week home-based flexibility exercise programme.

DETAILED DESCRIPTION:
Regular resistance training can lead to a variety of health benefits including increases in muscle size and strength, reductions on body fat, increased metabolic rate, glycaemic control, decreased blood pressure and improved blood lipid profiles. Because of this, current physical activity guidelines recommend undertaking muscle strengthening activities involving major muscle groups two days a week or more, alongside at least 150 minutes per week of moderate intensity physical activity (or 75 minutes per week of vigorous intensity physical activity). However, only small portion of the population achieves the muscle strengthening aspect of the guidelines.

Why participation in muscle-strengthening exercise is low is not clear but people identify several barriers including the lack of time, the effort involved, lack of purpose, pain due to injury, negative experiences of prescriptive exercise, apathy, illness, injury inclement weather and work commitment. In addition, some women have expressed a worry of looking 'manly' or 'bulking up' if they undertake resistance exercise. A further potential barrier is lack of access to a gym with appropriate equipment to perform resistance exercise, or dislike of a gym setting. Thus, identifying approaches to find a safe, enjoyable and accessible programme that minimises the burden of performing resistance exercise, and identifying a minimal amount of resistance training which can provide benefits is a key issue which could help more people to undertake muscle strengthening exercises.

Meta-analyses indicate that while performing resistance exercise two or more times per week of resistance exercise per muscle group appears to be optimal to maximise strength gains, a single set of resistance exercise per muscle group per week, if performed to failure is sufficient to induce substantial strength changes.

The main aim of this study is to compare the effects of an app-based home-based resistance exercise programme vs a home-based flexibility programme on muscular endurance (number of press-ups, time achieved in half-squat test, and time achieved in plank test, assessed online during a zoom call) and flexibility (sit and reach, assessed online during a zoom call) in healthy adults. Secondary aims are a) to determine participants' adherence to both exercise programmes, b) to determine participants' choice of weekly exercise volume (compared to minimum prescription) in both exercise programmes c) to determine participants' distribution of exercise throughout the week in both exercise programmes d) to determine the effects of a exercise programmes on well-being, and finally e) to determine participants' perceptions, feelings, thoughts, enjoyment, tolerance and acceptability of both exercise programmes.

The study is a randomized control trial in which the flexibility exercise group will undergo a 12-week home-based flexibility exercise programme. The resistance exercise group will undergo a 12-week home-based resistance exercise programme. Participants will be asked to perform a minimum amount of resistance or flexibility exercise of 1 set/week for each of six exercises and will have the opportunity to increase their volume of exercise to 2 sets or 3 sets/week per exercise if it is their choice. In addition, participants will be able to distribute the exercises during the week according to their preference (all in one day or spread over several days of the week, etc.). Participants will be encouraged to have a minimum of one day of rest per week.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years old.
* Perform 30 minutes or more of aerobic vigorous physical activity per week.
* Do not to perform any kind of resistance exercise.

Exclusion Criteria:

* Failure of the Physical Activity Readiness Questionnaire Plus (PAR-Q+)
* Perform 30 minutes or more of vigorous intensity exercise from the International Physical Activity Questionnaire (IPAQ)
* To have a job that compromises manual labour
* History of cardiovascular disease
* Diabetes
* Any other illness that would prevent the participation in a resistance exercise or flexibility exercise programme.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-12-06 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of press ups | 0 -12 weeks
  Change in number of press ups

SECONDARY OUTCOMES:
Number of press-ups | 0-6 weeks
  Change in the number of press ups
Number of press-ups | 6-12 weeks
  Change in the number of press ups
Time holding half-squat position | 0-12 weeks
  Change in the time holding half squat position
Time holding half-squat position | 0-6 weeks
  Change in the time holding half squat position
Time holding half-squat position | 6-12 weeks
  Change in the time holding half squat position
Time holding plank position | 0-12 weeks
  Change in the time holding plank position
Time holding plank position | 0-6 weeks
  Change in the time holding plank position
Time holding plank position | 6-12 weeks
  Change in the time holding plank position
Distance achieved in the sit-and-reach test | 0-12 weeks
  Change in distance achieved in the sit-and-reach test
Distance achieved in the sit-and-reach test | 0-6 weeks
  Change in distance achieved in the sit-and-reach test
Distance achieved in the sit-and-reach test | 6-12 weeks
  Change in distance achieved in the sit-and-reach test

CONTACTS AND LOCATIONS:
Overall Officials: Jason Gill, PhD, Principal Investigator — University of Glasgow
Locations (1):
- University of Glasgow, Glasgow, United Kingdom